CLINICAL TRIAL: NCT03823638
Title: A Phase II Single Center, Randomized, Double Blind and Placebo Controlled Study Assessing the Safety, Tolerability and Effects of Progressively Increased Dose of Oral Mannitol in Parkinson's Disease
Brief Title: Safety, Tolerability and Effects of Mannitol in Parkinson's Disease
Acronym: PD-mannitol
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, ARKADIR DAVID, Principal Investigator, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0346-17-HMO-CTIL
Record Dates: First submitted 2018-11-20; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-Mannitol (Experimental): Oral Supplement of the investigated substance: D-Mannitol powder (manufacturer Roquette)
  Interventions: Dietary Supplement: Oral D-Mannitol of Placebo
- Placebo (Placebo Comparator): Oral Supplement of the placebo: Dextrose monohydrate powder (manufacturer Roquette)
  Interventions: Dietary Supplement: Oral D-Mannitol of Placebo

INTERVENTIONS:
Dietary Supplement: Oral D-Mannitol of Placebo — Gradually increased doses of oral D-Mannitol of Placebo (Dextrose monohydrate)

SUMMARY:
Parkinson's disease is a progressive neurodegenerative disease that causes disabling motor and cognitive impairments. Currently, no disease-modifying therapy exists for this disease. Mannitol, a naturally-occurring substance, which is commonly used as sweetener, was offered as such agent. In this phase II, safety, tolerability-based dose finding, and efficacy study, mannitol or placebo (dextrose) in escalating doses will be given to patients with Parkinson's disease for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and signing of informed consent form.
2. Age 40-75 years at the day of visit 1.
3. Diagnosis of Parkinson's disease that is based on the United Kingdom brain bank criteria diagnosed after the age of 40.
4. Stable regime of anti-parkinsonian medication for at least 4 weeks at the day of visit 1.

Exclusion Criteria:

1. Patients with motor deficits that require administration of symptomatic therapy more than 4 times per day at the day of visit 1.
2. Patients on advanced therapy for Parkinson's disease (sub-cutaneous apomorphine, deep brain stimulation or intra-jejunal levodopa infusion).
3. Patients with dementia reflected by a Mini-mental state examination (MoCA) ≥ 24.
4. Patient with legal guardian.
5. History of psychosis or use of dopamine receptor blocking agent on the year proceeding at the visit 1. Quetiapine at dose lower or equal 50 mg per day prescribed for indication other than psychosis is allowed.
6. Suspected Parkinsonian syndrome other than Parkinson's disease.
7. Use of medical marihuana on the month proceeding visit 1.
8. Pregnant or lactating women, or fertile woman who does not use contraceptive. Woman of child-bearing potential must have a negative urine Human chorionic gonadotropin (hCG) and will be monitored by repeated urine tests.
9. Patient with significantly impaired renal functions (urea or creatinine values 20% above the upper norm limit).
10. Diabetes mellitus.
11. Clinical evidence for congestive heart failure.
12. Patient with symptomatic orthostatic hypotension.
13. Based on investigator's opinion, any medical condition that may progress due to consumption of oral mannitol or glucose.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of oral mannitol in Parkinson's disease as assessed by the number of mannitol-related adverse events, clinically significant changes in vital signs and clinically significant abnormalities in laboratory results. | 36 weeks
  Safety will be assessed by the number of treatment-related adverse events, number of patients with clinically significant change of vital signs (supine and standing blood pressure and pulse) and number of patients with clinically significant change in laboratory results (electrolytes, renal and liver functions, blood count).
Tolerability of oral mannitol in Parkinson's disease as assessed by the maximal daily dose (in grams) of mannitol that does not cause discomfort. | 36 weeks
  Tolerability of oral mannitol in Parkinson's disease as assessed by the maximal daily dose (in grams, up to 18 grams per day) of mannitol that does not cause discomfort based on the subjective report by the patient.

SECONDARY OUTCOMES:
Time-interval for starting symptomatic therapy (in days) between baseline and week 36, in patients not receiving symptomatic therapy at baseline. | 36 weeks
  Median time interval will be reported. P-Values as assessed by Mann-Whitney test will be reported. Longer time interval will be considered as a better outcome.
Change in levodopa-equivalent dose units between baseline and week 36. | 36 weeks
  Total levodopa-equivalent dose (LED units) will be calculated based on Tomlinson, Mov Disord 2010. P-Values as assessed by Mann-Whitney test will be reported. Smaller change will be considered as a better outcome.
Change of Brief Smell Identification Test (B-SIT) score between baseline and week 36. | 36 weeks
  Median and range of change will be reported. P-Values as assessed by Mann-Whitney test will be reported. Higher absolute positive value (reflecting improved smell) or lower absolute negative value (slower deterioration) will be considered as better outcomes.
Change in constipation assesment (CAS) score between baseline and week 36. | 36 weeks
  Median and range of change will be reported. Change in score will be reported. P-Values as assessed by Mann-Whitney test will be reported. Lower absolute positive value or higher absolute negative value will be considered as better outcomes.
Change in Montreal Cognitive Assessment (MoCA) test score between baseline and week 36. | 36 weeks
  P-Values as assessed by Mann-Whitney test will be reported. Higher absolute positive value or lower absolute negative value will be considered as better outcomes.
Change in non-motor symptoms of Parkinson's disease scale (NMSS) between baseline and week 36. | 36 weeks
  Median and range of change will be reported. P-Values as assessed by Mann-Whitney test will be reported. Lower absolute positive value or higher absolute negative value will be considered as better outcomes.
Change in the ratio of total-to-proteinase K-resistant α-synuclein in red blood cells (RBC) measured by enzyme-linked immunosorbent assay (ELISA)between baseline and week 36. | 36 weeks
  Median and range of change will be reported. P-Values as assessed by Mann-Whitney test will be reported. Higher absolute positive value or lower absolute negative value will be considered as better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No